CLINICAL TRIAL: NCT06972914
Title: Effect of Different Wearing Duration of Braces on Short-term Functional Recovery After Anterior Cruciate Ligament Reconstruction
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024001
Record Dates: First submitted 2025-04-29; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: Anterior cruciate ligament reconstruction; rehabilitation; brace

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Age, sex, time of onset, diagnosis, underlying disease, complications, perioperative status, knee circumference, Lysholm score, IKDC score, muscle strength, graft maturity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the correlation between wearing time of different braces and short-term functional changes such as knee functional score, knee circumference and postoperative recovery Angle after ACL reconstruction, and provide preliminary evidence and key data for subsequent research on whether and how long it is necessary to wear braces after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

-Patients with acute anterior cruciate ligament injury undergoing anterior cruciate ligament reconstruction

Exclusion Criteria:

-Refused to sign the informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after anterior cruciate ligament reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Thigh circumference | Preoperative, postoperative 3 weeks, 6 weeks, 3 months, 6 months, 9 months
  Thigh dimension: centimeters(cm)
Degree of Joint range of motion | Preoperative, postoperative 3 weeks, 6 weeks, 3 months, 6 months, 9 months
  Degree of Joint range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital of Chongli, Chongli, Hebei, China